CLINICAL TRIAL: NCT04952857
Title: Short Term, High Dose Vitamin D Supplementation in Moderate to Severe COVID-19 Disease
Acronym: SHADE-S
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Ashu Rastogi, Associate Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INT/2020/001068
Record Dates: First submitted 2021-06-08; First posted 2021-07-07 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Vitamn D 6 lakh IU oral stat
  Interventions: Drug: cholecalciferol 6 lakh IU
- Placebo (Placebo Comparator): Placebo equal volume/ weight
  Interventions: Drug: cholecalciferol 6 lakh IU

INTERVENTIONS:
Drug: cholecalciferol 6 lakh IU — vitamin D levels and serum calcium will be assessed at day 3,7, 14.
  Other Names: vitamin D

SUMMARY:
COVID-19 caused by SARS-CoV-2 virus has affected the lives of millions of individuals globally and also severely strained the medical community. Pre-symptomatic and asymptomatic SARS-CoV-2 positive individuals far outnumber the symptomatic ones or those with severe disease. The transmission potential of SARS CoV-2 is potentially greater than earlier viral outbreaks of SARS-CoV and MERS-CoV.Routine measures of social distancing, personal hand hygiene and limited outdoor contact activities have shown benefits to limit corona virus infection. However, the role of vitamin D in SARS-CoV-2 infection is sparingly explored despite the knowledge of an immunomodulatory role and protective effect of vitamin D against viral infections. Meta-analysis of five clinical trials of vitamin D supplementation found that those receiving vitamin D supplementation had fewer respiratory tract infections (odds ratio = 0.58 (95%CI, 0.42 - 0.81).Any immune-modulatory effect of vitamin D is likely to be observed at levels which are considered higher than that required for normal bone metabolism.

ELIGIBILITY:
Inclusion Criteria:

1. RT-PCR proven SARS-CoV-2 infection or computed tomography scan findings compatible with the COVID19 disease (bilateral multifocal ground-glass opacities ≥50%)
2. Moderate to severe COVID-19 defined by PFR ratio of <200
3. SOFA score>4
4. Patients with vitamin D deficiency defined as 25 (OH)D level<20 ng/ml
5. Age>18 years

Exclusion Criteria:

* 1. Vitamin D sufficient or already receiving vitamin D supplements 2. Active malignancy 3. Hypercalcemia, hyperparathyroidism 4. Chronic kidney disease (eGFR<30 ml/min) 5. Pregnant and lactating women 6. Patient on mechanical ventilation at ICU admission

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Sequential Organ Failure Assessment (SOFA) | 7 days
  Sequential Organ Failure Assessment score at day 7. SOFA score range from 1 to a maximum of 24. A greator score suggests worse outcome.

SECONDARY OUTCOMES:
Sequential Organ Failure Assessment (SOFA) Score | 3 days
  Sequential Organ Failure Assessment score at day 3. SOFA score range from 1 to a maximum of 24. A greator score suggests worse outcome.
Sequential Organ Failure Assessment (SOFA) score | 14 days
  Sequential Organ Failure Assessment (SOFA) score at day 14. SOFA score range from 1 to a maximum of 24 score. A greator score suggests worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Deptt of Endocrinology, Chandigarh, India

REFERENCES:
- [Derived] Singh A, Rastogi A, Puri GD, Ganesh V, Naik NB, Kajal K, Kahlon S, Soni SL, Kaloria N, Saini K, Hazarika A, Mahajan V, Singla K, Bhadada S, Soni V. Therapeutic high-dose vitamin D for vitamin D-deficient severe COVID-19 disease: randomized, double-blind, placebo-controlled study (SHADE-S). J Public Health (Oxf). 2024 May 29;46(2):256-266. doi: 10.1093/pubmed/fdae007. PMID 38291897